CLINICAL TRIAL: NCT02558946
Title: Perioperative Pelvic Floor Muscle Training May Improve Recovery of Continence in Men with Localized Prostate Cancer Undergoing Robot-Assisted Radical Prostatectomy
Brief Title: Physical Therapy for Men Undergoing Prostatectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Indiana University Health (Other)
Responsible Party: Principal Investigator, Ronald Boris, Associate Professor, Urology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1501440753
Record Dates: First submitted 2015-09-18; First posted 2015-09-24 (Estimated); Last update posted 2024-11-04 (Actual); Status verified 2024-07

CONDITIONS: Prostate Cancer; Urinary Incontinence; Pelvic Floor Physical Therapy
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Incontinence | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical Therapy Treatment Group (Active Comparator): Written and verbal information on performing Kegel exercises (exercises that aim to strengthen pelvic floor muscles) will be provided at the pre-op clinic visit. The treatment group will receive pelvic floor muscle training through a course of three one-hour sessions with a trained pelvic floor physical therapist in addition to the current standard information from their surgeon. The physical therapy sessions will be conducted at 1-6 weeks preoperative, 7-10 days postoperative, and 4-8 weeks postoperative .
  Interventions: Behavioral: Pelvic Floor Muscle Physical Therapy
- Control Group (Active Comparator): Written and verbal information on performing Kegel exercises (exercises that aim to strengthen pelvic floor muscles) will be provided at the pre-op clinic visit.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Pelvic Floor Muscle Physical Therapy — The treatment group will receive pelvic floor muscle training through a course of three one-hour sessions with a trained pelvic floor physical therapist in addition to the current standard information from their surgeon. The physical therapy sessions will be conducted at 1-6 weeks preoperative, 1 week postoperative, and 4-6 weeks postoperative and will be coordinated with surgeon appointments to minimize any inconvenience and travel time.
  Arms: Physical Therapy Treatment Group
Behavioral: Control Group — At the cancer consultation visit, subjects will be educated by the urologist or urology team member regarding surgical and postoperative expectations. At this time, subjects will be provided verbal instruction and written information regarding Kegel exercises. Subjects in the control group may decide the duration and frequency of home exercise performance.
  Arms: Control Group

SUMMARY:
The purpose of this study is to determine if pelvic floor muscle training with a physical therapist before and after surgery will improve health-related quality of life following robot-assisted radical prostatectomy.

DETAILED DESCRIPTION:
Goals of the present study will be to determine whether initiating pelvic floor muscle training preoperatively improves quality of life symptoms related specifically to urinary health following robot-assisted radical prostatectomy. Drawing definitive conclusions from past studies is challenging secondary to various inconsistencies including: variability of physical therapy intervention, poorly defined definitions of continence, as well as poorly defined quality of life measurements. Additionally, the vast majority of studies combined open and robotic prostatectomy increasing cohort heterogeneity and further blurring interpretation of results. The investigators' study will focus exclusively on patients undergoing robot-assisted radical prostatectomy. Standardized pelvic floor muscle therapy as well as clearly defined patient outcomes (ie: validated questionnaires) will be utilized to determine whether preoperative initiation of formal pelvic floor physical therapy can improve health-related quality of life following surgery.

In the era of robot-assisted radical prostatectomy does physical therapist initiated preoperative pelvic floor muscle training lessen the expected postoperative drop off in urinary related quality of life and/or improve patient's recovery of continence following surgery?

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduling to undergo robot-assisted radical prostatectomy
* Patients willing and able to complete the EPIC questionnaire in its entirety
* Ability to provide informed consent

Exclusion Criteria:

* Previous prostate surgery
* Radiation treatment
* History of incontinence defined as any pad use for urinary leakage in the past 6 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2015-06-29 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
• Comparison of post-op EPIC scores in the two study groups | 4 to 8 weeks post-op

SECONDARY OUTCOMES:
Return to continence following surgery | Up to 12 months post-op

CONTACTS AND LOCATIONS:
Locations (1):
- IU Health Methodist Hospital and IU Health University Hospital, Indianapolis, Indiana, United States